CLINICAL TRIAL: NCT01172847
Title: An Open-label, Multiple Dose, Randomized, Three-period Crossover Study in Healthy Subjects to Evaluate the Effect of Co-administration of Oseltamivir (Ro 64-0796) 75 mg Twice Daily and Rimantadine 100 mg Twice Daily on the Pharmacokinetic Properties of Oseltamivir and Rimantadine.
Brief Title: A Pharmacokinetic Study on Co-administration of Tamiflu (Oseltamivir) and Rimantadine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP22770; 2009-012742-23
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Oseltamivir; Rimantadine

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: oseltamivir [Tamiflu]
- B (Active Comparator)
  Interventions: Drug: rimantadine
- C (Experimental)
  Interventions: Drug: oseltamivir [Tamiflu]; Drug: rimantadine

INTERVENTIONS:
Drug: oseltamivir [Tamiflu] — multiple oral doses
  Arms: A; C
Drug: rimantadine — multiple oral doses
  Arms: B; C

SUMMARY:
This open label, randomized, three-period crossover study will evaluate the effect of co-administration of Tamiflu (oseltamivir) and rimantadine on the pharmacokinetics of Tamiflu and rimantadine. Healthy volunteers will receive multiple oral doses of Tamiflu, rimantadine or Tamiflu plus rimantadine in random order, with a minimum wash-out period of 7 days between treatments. Anticipated time on study is up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18 to 45 years
* Healthy as judged by general physical examination, medical history, vital signs, 12-lead ECG and laboratory tests
* Body Mass Index (BMI) 18-34 kg/m2
* Willing not to participate in any other trial including an investigational drug for 3 months following the last dose
* Male subjects must agree to use a barrier contraception during the study and for 3 months after discontinuation of treatment
* Female subjects of non-child bearing potential or under effective contraception who are either post-menopausal, surgically sterile, or who agree to use barrier contraception during the whole study in addition to an intrauterine device or hormonal contraception for at least 3 months prior to 1st dose, during the study and for 3 months after discontinuation of treatment

Exclusion Criteria:

* History of or current clinically significant disease or disorder
* Positive Hepatitis B, Hepatitis C, HIV 1 or 2 test result
* Positive pregnancy test or lactating women
* Clinically relevant history of allergy or hypersensitivity
* Clinically relevant history of abuse of alcohol or other drugs; tobacco smoking is allowed (</= 10 cigarettes a day or equivalent of tobacco in cigars or pipe)
* Any major illness within 30 days prior to screening examination
* Administration of any medication during the 7 days prior to drug administration, except for paracetamol and aspirin (up to 48 hours before first dose) and oral contraceptives
* Participation in a clinical study with an investigational drug within 3 months prior to study day 1
* Donation or loss of more than 500 mL of blood within the 3 months prior to study day 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States from 04 August 2009 to 28 September 2009. A total of 40 participants were screened.
Pre-assignment Details: Of 40 participants, 24 participants were enrolled.
Groups:
- Oseltamivir; Rimantadine; Oseltamivir + Rimantadine: Participants received treatments in 3 periods as: Oseltamivir 75 milligram [mg] (twice a day orally for 5 days), Rimantadine 100 mg (twice a day orally for 5 days), and Oseltamivir 75 mg + Rimantadine 100 mg (twice a day orally for 5 days) in a randomly determined sequence with a minimum 7-day wash out period between consecutive treatments periods.
Period: Overall Study
Arm/Group | Oseltamivir; Rimantadine; Oseltamivir + Rimantadine
Started | 24
Oseltamivir | 24
Rimantadine | 22
Oseltamivir + Rimantadine | 21
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oseltamivir; Rimantadine; Oseltamivir + Rimantadine
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Steady State Area Under the Plasma Concentration Versus Time Curve From 0 to 12 Hours After Dosing (AUC0-12) of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. AUC0-12 of oseltamivir and oseltamivir carboxylate were calculated following the administration of oseltamivir alone or in combination with rimantadine, using the linear trapezoidal rule.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 5
Population: Pharmacokinetics (PK) analysis population included all participants who were adhered to the protocol.
Measure: Least Squares Mean (90% Confidence Interval); unit: hours (h)*nanogram (ng)/milliliter (mL)
Groups:
- Oseltamivir: Participants received oseltamivir 75 mg twice a day orally for 5 days.
- Oseltamivir + Rimantadine: Participants received oseltamivir 75 mg + rimantadine 100 mg twice a day orally for 5 days.
Arm/Group | Oseltamivir | Oseltamivir + Rimantadine
Number analyzed (Participants) | 21 | 21
hours (h)*nanogram (ng)/milliliter (mL)
  Oseltamivir | 5.092 [5.041 to 5.143] | 5.070 [5.019 to 5.121]
  Oseltamivir Carboxylate | 8.008 [7.982 to 8.034] | 7.990 [7.964 to 8.017]
Statistical Analysis 1: Comparison: Oseltamivir vs Oseltamivir + Rimantadine; Mean exposure ratio of oseltamivir; Test type: Superiority or Other; mean exposure ratio = 0.98, 90% CI 2-sided [0.91 to 1.05] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model
Statistical Analysis 2: Comparison: Oseltamivir; Mean exposure ratio of oseltamivir carboxylate; Test type: Superiority or Other; mean exposure ratio = 0.98, 90% CI 2-sided [0.95 to 1.02] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model

2. Primary Outcome: Steady State Area Under the Plasma Concentration Versus Time Curve From 0 to 12 Hours After Dosing (AUC0-12) of Rimantadine
Description: AUC0-12 of rimantadine was calculated following the administration of rimantadine alone or in combination with oseltamivir, using the linear trapezoidal rule.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 5
Population: Pharmacokinetic analysis population included all participants who were adhered to the protocol.
Measure: Least Squares Mean (90% Confidence Interval); unit: h*ng/mL
Groups:
- Rimantadine; Oseltamivir + Rimantadine: Participants received oseltamivir 75 mg + rimantadine 100 mg twice a day orally for 5 days.
Arm/Group | Rimantadine | Oseltamivir + Rimantadine
Number analyzed (Participants) | 21 | 21
h*ng/mL | 8.371 [8.349 to 8.394] | 8.398 [8.376 to 8.421]
Statistical Analysis 1: Comparison: Rimantadine vs Oseltamivir + Rimantadine; Mean exposure ratio of rimantadine; Test type: Superiority or Other; mean exposure ratio = 1.03, 90% CI 2-sided [1.00 to 1.06] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. Cmax of oseltamivir and oseltamivir carboxylate were calculated following the administration of oseltamivir alone or in combination with rimantadine and was directly observed from the data.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 5
Population: PK analysis population included all participants who were adhered to the protocol.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Oseltamivir | Oseltamivir + Rimantadine
Number analyzed (Participants) | 21 | 21
ng/mL
  Oseltamivir | 4.395 [4.317 to 4.472] | 4.249 [4.171 to 4.326]
  Oseltamivir Carboxylate | 5.940 [5.894 to 5.986] | 5.921 [5.874 to 5.967]
Statistical Analysis 1: Comparison: Oseltamivir vs Oseltamivir + Rimantadine; Mean exposure ratio of oseltamivir; Test type: Superiority or Other; mean exposure ratio = 0.86, 90% CI 2-sided [0.77 to 0.96] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model
Statistical Analysis 2: Comparison: Oseltamivir vs Oseltamivir + Rimantadine; Mean exposure ratio of oseltamivir carboxylate; Test type: Superiority or Other; mean exposure ratio = 0.98, 90% CI 2-sided [0.92 to 1.05] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Rimantadine
Description: Cmax of rimantadine was calculated following the administration of rimantadine alone or in combination with oseltamivir and was directly observed from the data.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 5
Population: PK analysis population included all participants who were adhered to the protocol.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Oseltamivir | Oseltamivir + Rimantadine
Number analyzed (Participants) | 21 | 21
ng/mL | 6.036 [6.010 to 6.061] | 6.062 [6.036 to 6.087]
Statistical Analysis 1: Comparison: Oseltamivir vs Oseltamivir + Rimantadine; mean exposure ratio of rimantadine; Test type: Superiority or Other; mean exposure ratio = 1.03, 90% CI 2-sided [0.99 to 1.06] — Estimate of the treatment difference and corresponding 90% CI was derived from the back-transformed model

5. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 11 weeks
Population: Safety Population included all participants who received at least one dose of the study medication, whether prematurely withdrawn from the study or not.
Measure: Number; unit: participants
Groups:
- Rimantadine: Participants received rimantadine 100 mg twice a day orally for 5 days.
Arm/Group | Oseltamivir | Rimantadine | Oseltamivir + Rimantadine
Number analyzed (Participants) | 24 | 22 | 21
participants | 8 | 6 | 4

6. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs included heart rate (HR), blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), and body temperature. Blood pressure and pulse rate were recorded when participants were rested in a supine position for at least 5 minutes and after standing for 2 minutes. Vital signs values that fall outside the investigator's normal ranges were recorded.
Time Frame: Screening (Days -28 to -2); pre-dose and 2h post-dose on D1 and D5 of each treatment period; at Follow-up visit (10 -14 days after last dose) for blood pressure and HR; Screening; Day -1 of each treatment period; Follow-up visit for temperature
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Oseltamivir | Rimantadine | Oseltamivir + Rimantadine
Number analyzed (Participants) | 24 | 22 | 21
participants
  High- SBP | 6 | 1 | 2
  High- DBP | 2 | 0 | 0
  High- DBP standing | 8 | 6 | 2
  High- SBP standing | 7 | 4 | 3
  High- HR | 2 | 0 | 0
  High- HR standing | 2 | 1 | 2
  Low- Temperature | 7 | 11 | 8

7. Secondary Outcome: Number of Participants With Marked Abnormality in Laboratory Parameters
Description: Laboratory analysis included hematology (hemoglobin, hematocrit, erythrocytes, platelets counts, leukocytes counts, neutrophils, eosinophils, lymphocytes, basophils, and monocytes);, biochemistry (aspartate aminotransferase , alanine aminotransferase, gamma glutamyl trans peptidase, total bilirubin, alkaline phosphatase, lactate dehydrogenase, albumin, creatinine, urea, creatine phosphokinase, total protein, sodium, chloride, calcium, phosphate, potassium, glucose (fasting), amylase, lipase, total cholesterol, and calculated creatinine clearance); and urinalysis.
  Marked laboratory test values (high and low) falling outside the marked reference range and which also represents a clinically relevant change from baseline of at least a designated amount were recoded. In this study, marked abnormality ranges for phosphate as 0.75 - 1.60 millimole (mmol)/L and proteinuria (0 to 4+, and 1).
Time Frame: Screening; Day -1 and Day 5 (pre-dose) of each treatment period; Follow-up visit
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Oseltamivir | Rimantadine | Oseltamivir + Rimantadine
Number analyzed (Participants) | 24 | 22 | 21
participants
  Phosphate High | 1 | 1 | 1
  Phosphate Low | 1 | 0 | 0
  Proteinuria | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant or Treatment Related Changes in Electrocardiogram (ECG)
Description: ECG was recorded when participants were rested in a supine position for at least 5 minutes.
Time Frame: Screening; pre-dose on Day 1 and Day 5 of each treatment period; Follow-up visit
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Oseltamivir | Rimantadine | Oseltamivir + Rimantadine
Number analyzed (Participants) | 24 | 22 | 21
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 11 weeks
Description: SAEs and other AEs were collected in the safety population which included all participants who received at least one dose of the study medication, whether prematurely withdrawn from the study or not.
Arm/Group | Oseltamivir | Rimantadine | Oseltamivir + Rimantadine
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 8/24 | 6/22 | 4/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir (N=24) | Rimantadine (N=22) | Oseltamivir + Rimantadine (N=21)
Toothache (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.